CLINICAL TRIAL: NCT01723852
Title: Vitamin D Intervention in Infants
Acronym: VIDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: The Finnish Governmental Special Subsidy for Health Sciences Research (Unknown); Päivikki and Sakari Sohlberg Foundation, Finland (Other); The Finnish Medical Association (Other)
Responsible Party: Principal Investigator, Sture Andersson, Professor of Neonatology, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VIDI-2012-01
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Vitamin D Status
Keywords: Vitamin D; Infectious diseases; cognitive development; Bone mineral density; Immunoregulation; Allergy; Growth
MeSH Terms: conditions — Communicable Diseases; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D supplement (Active Comparator): Vitamin D supplement according to national guidelines (10 ug/day) from 2 weeks to 2 years of age
  Interventions: Dietary Supplement: Vitamin D at 10 ug/day
- Vitamin D supplement at 30 ug/day (Active Comparator): Vitamin D supplement at 30 ug/day from 2 weeks to 2 years of age
  Interventions: Dietary Supplement: Vitamin D at 30 ug/day

INTERVENTIONS:
Dietary Supplement: Vitamin D at 30 ug/day
  Arms: Vitamin D supplement at 30 ug/day
Dietary Supplement: Vitamin D at 10 ug/day
  Arms: Vitamin D supplement

SUMMARY:
The study is a randomized, controlled, double blinded study evaluating the effect of recommended (400 IU) and 1 200 IU daily vitamin D substitution, given from 2 weeks to 2 years of age, on growth, bone development, neurologic and cognitive development, frequence of infectious diseases, allergic symptoms, and development of immunoregulation assessed at 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at term (37-42 wks, weight appropriate for gestational age) are included in the study

Exclusion Criteria:

* Non Caucasian mother
* Any continuous regular medication of mother
* Treatment at neonatal intensive care unit
* Antibiotic treatment of the infant
* Congenital malformations of the newborn
* Treatment with ventilation support (continuous nasal positive airway pressure) for over 24 hours
* Glucose infusion of the newborn
* Neurological symptoms of the newborn
* Phototherapy for jaundice of the newborn
* Need for nasogastric feeding of the newborn

Max Age: 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Growth | 2 years of age
  Measurement of growth at 2 years of age
Neurologic and cognitive development | At 2 years of age
  By means of questionnaires and, on a randomly selected group of study subjects, cognitive function testing to assess neurologic and cognitive development
Frequency of allergic symptoms and infection | At 2 years of age
  Assessment of the frequency of allergic symptoms and infections by means of questionnaires, hospital discharge records and prescription data.
Development of immunoregulation | At 2 years of age
  Assessment of the tolerogenic properties of T-cells and dendritic cell function from blood sample in a subgroup of 100 study subjects.
Bone mineral density | 2 years of age
  Bone mineral density is measured by dual energy x-ray absorptiometry and peripheral quantitative computerized tomography

CONTACTS AND LOCATIONS:
Overall Officials: Sture Andersson, MD, PhD, Principal Investigator — Helsinki University Central Hospital, Children's Hospital
Locations (1):
- Kätilöopisto Maternity Hospital, Helsinki, Finland

REFERENCES:
- [Background] Holmlund-Suila E, Viljakainen H, Hytinantti T, Lamberg-Allardt C, Andersson S, Makitie O. High-dose vitamin d intervention in infants--effects on vitamin d status, calcium homeostasis, and bone strength. J Clin Endocrinol Metab. 2012 Nov;97(11):4139-47. doi: 10.1210/jc.2012-1575. Epub 2012 Aug 29. PMID 22933541
- [Background] Helve O, Viljakainen H, Holmlund-Suila E, Rosendahl J, Hauta-Alus H, Enlund-Cerullo M, Valkama S, Heinonen K, Raikkonen K, Hytinantti T, Makitie O, Andersson S. Towards evidence-based vitamin D supplementation in infants: vitamin D intervention in infants (VIDI) - study design and methods of a randomised controlled double-blinded intervention study. BMC Pediatr. 2017 Mar 29;17(1):91. doi: 10.1186/s12887-017-0845-5. PMID 28356142
- [Result] Rosendahl J, Holmlund-Suila E, Helve O, Viljakainen H, Hauta-Alus H, Valkama S, Enlund-Cerullo M, Hytinantti T, Tervahartiala T, Sorsa T, Makitie O, Andersson S. 25-hydroxyvitamin D correlates with inflammatory markers in cord blood of healthy newborns. Pediatr Res. 2017 May;81(5):731-735. doi: 10.1038/pr.2017.9. Epub 2017 Jan 13. PMID 28085793
- [Result] Hauta-Alus HH, Holmlund-Suila EM, Rita HJ, Enlund-Cerullo M, Rosendahl J, Valkama SM, Helve OM, Hytinantti TK, Surcel HM, Makitie OM, Andersson S, Viljakainen HT. Season, dietary factors, and physical activity modify 25-hydroxyvitamin D concentration during pregnancy. Eur J Nutr. 2018 Jun;57(4):1369-1379. doi: 10.1007/s00394-017-1417-z. Epub 2017 Mar 2. PMID 28255653
- [Result] Valkama S, Holmlund-Suila E, Enlund-Cerullo M, Rosendahl J, Hauta-Alus H, Helve O, Hytinantti T, Viljakainen H, Andersson S, Makitie O. No Severe Hypercalcemia with Daily Vitamin D3 Supplementation of up to 30 microg during the First Year of Life. Horm Res Paediatr. 2017;88(2):147-154. doi: 10.1159/000477298. Epub 2017 Jun 23. PMID 28647736
- [Result] Holmlund-Suila E, Enlund-Cerullo M, Valkama S, Hauta-Alus H, Rosendahl J, Helve O, Hytinantti T, Viljakainen H, Andersson S, Makitie O. Sex and Iron Modify Fibroblast Growth Factor 23 Concentration in 1-Year-Old Children. J Clin Endocrinol Metab. 2017 Dec 1;102(12):4526-4533. doi: 10.1210/jc.2017-01211. PMID 29029193
- [Derived] Seppala V, Sandboge S, Holmlund-Suila E, Hauta-Alus H, Lintula S, Kajantie E, Makitie O, Andersson S, Raikkonen K, Heinonen K. Early life vitamin D and neurocognitive abilities at age 6-8 years: a randomized clinical trial and observational analysis. Eur Child Adolesc Psychiatry. 2025 Oct 10. doi: 10.1007/s00787-025-02891-7. Online ahead of print. PMID 41071326
- [Derived] Enlund-Cerullo M, Holmlund-Suila E, Valkama S, Hauta-Alus H, Rosendahl J, Andersson S, Pekkinen M, Makitie O. Variation in the fibroblast growth factor 23 (FGF23) gene associates with serum FGF23 and bone strength in infants. Front Genet. 2023 May 22;14:1192368. doi: 10.3389/fgene.2023.1192368. eCollection 2023. PMID 37284066
- [Derived] Sandboge S, Raikkonen K, Lahti-Pulkkinen M, Hauta-Alus H, Holmlund-Suila E, Girchenko P, Kajantie E, Makitie O, Andersson S, Heinonen K. Effect of Vitamin D3 Supplementation in the First 2 Years of Life on Psychiatric Symptoms at Ages 6 to 8 Years: A Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2314319. doi: 10.1001/jamanetworkopen.2023.14319. PMID 37204794
- [Derived] Pontan F, Hauta-Alus H, Valkama S, Rosendahl J, Enlund-Cerullo M, Andersson S, Makitie O, Holmlund-Suila E. Alkaline Phosphatase and Hyperphosphatasemia in Vitamin D Trial in Healthy Infants and Toddlers. J Clin Endocrinol Metab. 2023 Sep 18;108(10):e1082-e1091. doi: 10.1210/clinem/dgad208. PMID 37061810
- [Derived] Holmlund-Suila EM, Hauta-Alus HH, Enlund-Cerullo M, Rosendahl J, Valkama SM, Andersson S, Makitie O. Iron status in early childhood is modified by diet, sex and growth: Secondary analysis of a randomized controlled vitamin D trial. Clin Nutr. 2022 Feb;41(2):279-287. doi: 10.1016/j.clnu.2021.12.013. Epub 2021 Dec 13. PMID 34999321
- [Derived] Tuovinen S, Raikkonen K, Holmlund-Suila E, Hauta-Alus H, Helve O, Rosendahl J, Enlund-Cerullo M, Kajantie E, Valkama S, Viljakainen H, Makitie O, Andersson S, Heinonen K. Effect of High-Dose vs Standard-Dose Vitamin D Supplementation on Neurodevelopment of Healthy Term Infants: A Randomized Clinical Trial. JAMA Netw Open. 2021 Sep 1;4(9):e2124493. doi: 10.1001/jamanetworkopen.2021.24493. PMID 34495336
- [Derived] Koljonen L, Enlund-Cerullo M, Hauta-Alus H, Holmlund-Suila E, Valkama S, Rosendahl J, Andersson S, Pekkinen M, Makitie O. Phosphate Concentrations and Modifying Factors in Healthy Children From 12 to 24 Months of Age. J Clin Endocrinol Metab. 2021 Sep 27;106(10):2865-2875. doi: 10.1210/clinem/dgab495. PMID 34214153
- [Derived] Hauta-Alus HH, Holmlund-Suila EM, Kajantie E, Rosendahl J, Valkama SM, Enlund-Cerullo M, Andersson S, Makitie O. The Effects of Vitamin D Supplementation During Infancy on Growth During the First 2 Years of Life. J Clin Endocrinol Metab. 2021 Mar 8;106(3):e1140-e1155. doi: 10.1210/clinem/dgaa943. PMID 33347567
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- [Derived] Valkama S, Holmlund-Suila E, Ireland A, Hauta-Alus H, Enlund-Cerullo M, Rosendahl J, Andersson S, Makitie O. Peripheral quantitative computed tomography (pQCT) in 12- and 24-month-old children - Practical aspects and descriptive data. Bone. 2020 Dec;141:115670. doi: 10.1016/j.bone.2020.115670. Epub 2020 Sep 30. PMID 33007527
- [Derived] Enlund-Cerullo M, Hauta-Alus H, Valkama S, Rosendahl J, Andersson S, Makitie O, Holmlund-Suila E. Fibroblast growth factor 23 concentrations and modifying factors in children from age 12 to 24 months. Bone. 2020 Dec;141:115629. doi: 10.1016/j.bone.2020.115629. Epub 2020 Sep 10. PMID 32919110
- [Derived] Enlund-Cerullo M, Koljonen L, Holmlund-Suila E, Hauta-Alus H, Rosendahl J, Valkama S, Helve O, Hytinantti T, Viljakainen H, Andersson S, Makitie O, Pekkinen M. Genetic Variation of the Vitamin D Binding Protein Affects Vitamin D Status and Response to Supplementation in Infants. J Clin Endocrinol Metab. 2019 Nov 1;104(11):5483-5498. doi: 10.1210/jc.2019-00630. PMID 31365099
- [Derived] Hauta-Alus HH, Kajantie E, Holmlund-Suila EM, Rosendahl J, Valkama SM, Enlund-Cerullo M, Helve OM, Hytinantti TK, Viljakainen H, Andersson S, Makitie O. High Pregnancy, Cord Blood, and Infant Vitamin D Concentrations May Predict Slower Infant Growth. J Clin Endocrinol Metab. 2019 Feb 1;104(2):397-407. doi: 10.1210/jc.2018-00602. PMID 30247704
- [Derived] Rosendahl J, Valkama S, Holmlund-Suila E, Enlund-Cerullo M, Hauta-Alus H, Helve O, Hytinantti T, Levalahti E, Kajantie E, Viljakainen H, Makitie O, Andersson S. Effect of Higher vs Standard Dosage of Vitamin D3 Supplementation on Bone Strength and Infection in Healthy Infants: A Randomized Clinical Trial. JAMA Pediatr. 2018 Jul 1;172(7):646-654. doi: 10.1001/jamapediatrics.2018.0602. PMID 29813149
- [Derived] Hauta-Alus HH, Viljakainen HT, Holmlund-Suila EM, Enlund-Cerullo M, Rosendahl J, Valkama SM, Helve OM, Hytinantti TK, Makitie OM, Andersson S. Maternal vitamin D status, gestational diabetes and infant birth size. BMC Pregnancy Childbirth. 2017 Dec 15;17(1):420. doi: 10.1186/s12884-017-1600-5. PMID 29246128